CLINICAL TRIAL: NCT02521753
Title: Effect Polyunsaturated Fatty Acids or Magnesium in Metabolic, Hormonal, and Inflammatory Profile in Obese Women With Polycystic Ovary Syndrome. A Randomized Clinical Trial
Brief Title: Omega 3 Polyunsaturated Fatty Acids (PUFA) or Magnesium in Obese Polycystic Ovary Syndrome Patients
Acronym: OMgObPCOS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It was not possible to continue recruiting due to SARSCov2 pandemia. Results obtained at that time were already published
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Mardia Guadalupe Lopez Alarcon, Investigador titular B, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2014-785-056
Record Dates: First submitted 2015-07-27; First posted 2015-08-13 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Polycystic Ovary Syndrome; Obesity
Keywords: Polycystic ovary syndrome; Obesity; Metformin; Magnesium; Polyunsaturated fatty acids
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity | interventions — Metformin; Magnesium; Docosahexaenoic Acids

STUDY DESIGN:
Masking Description: The study is open label. No blindness for participant or investigator is used
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metformin (Active Comparator): Metformin 850mg twice a day for six months
  Interventions: Drug: Metformin
- Magnesium (Experimental): Magnesium chloride 250mg daily for six months
  Interventions: Dietary Supplement: Magnesium
- PUFA omega 3 (Experimental): Eicosapentaenoic acid (EPA) + Docosahexaenoic acid (DHA) 1.1mg daily for six months
  Interventions: Dietary Supplement: PUFA

INTERVENTIONS:
Drug: Metformin — Intervention also includes weight reduction diet and exercise therapy
  Other Names: Glucophage
  Arms: Metformin
Dietary Supplement: Magnesium — Intervention also includes weight reduction diet and exercise therapy
  Other Names: Nature made magnesium
  Arms: Magnesium
Dietary Supplement: PUFA — Intervention also includes weight reduction diet and exercise therapy
  Other Names: Omega 3
  Arms: PUFA omega 3

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most prevalent endocrine disorder in reproductive age women. PCOS is usually characterized by an excessive androgen production, menstrual irregularities, and polycystic ovaries. Women with PCOS are often obese and have a varying degree of insulin resistance (IR). Weight reduction constitutes the initial treatment for these patients. Metformin has proven to be useful in IR and is frequently used in PCOS. However metformin use may be accompanied by gastrointestinal discomfort, and a high abandon rate. Other therapeutic alternatives such as magnesium and polyunsaturated fatty acids have been used in other IR states and may be useful in PCOS. The aim of this study is to asses the efficacy of these alternatives in obese PCOS patients.

DETAILED DESCRIPTION:
Polycystic Ovary Syndrome (PCOS)

ELIGIBILITY:
Inclusion Criteria:

* Polycystic Ovary Syndrome according to Rotterdam criteria,
* BMI ≥ 27 Kg/m2

Exclusion Criteria:

* Type 2 diabetes mellitus,
* in treatment for polycystic ovary syndrome features

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2025-03 (Actual)

PRIMARY OUTCOMES:
Metabolic profile | Six months after intervention
  Serum concentration of metabolic biomarkers (glucose, insulin, triglycerides, cholesterol, HDL, M and M/I value derived from a euglycemic clamp)

SECONDARY OUTCOMES:
Hormonal profile | Six months after intervention
  Serum concentration of hormones [Testosterone, dehydroepiandrosterone sulphate (DHEAs), sex hormone-binding globulin (SHBG), free androgen index (FAI)]

CONTACTS AND LOCATIONS:
Overall Officials: Mardia Guadalupe López Alarcón, MD, phD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Hospital de Gineco Obstetricia Centro Médico "La Raza", Mexico City, D.F., Mexico

IPD SHARING:
Plan to Share IPD: No
There is not a plan to share data